### Impact of Unexpected Death in Simulation: Skill Retention, Stress and Emotions

## **Data Analysis Plan**

**Primary Outcome:** Difference in retention of non-technical crisis resource management (CRM) skills using Ottawa Global Rating Scale (OGRS)

#### ANCOVA:

- Dependent variable: OGRS score (total score)
- Independent variable: Death vs. survival
- Covariates: Junior vs. senior; Acute vs. non-acute

## **Secondary Outcome 1**: Technical CRM skills (according to checklist)

 Same Videos to be provided for primary outcome will be scored using the "Task-specific checklist" (derived from American Heart Association's Megacode Checklist) and given a score out of 18

#### ANCOVA:

- Dependent variable: Task-specific checklist score (total score)
- Independent variable: Death vs. survival
- Covariates: Junior vs. senior; Acute vs. non-acute

## Secondary Outcome 2: Stress

## Measure 1: Salivary cortisol

Five time points (minutes passed since baseline):

- 1. Baseline (0 minutes) during the accommodation period at the beginning of the day
- 2. Before scenario (10 minutes)
- 3. Immediately after scenario (30 minutes)
- 4. 30 minutes after start of scenario (45 minutes)
- 5. After debrief (50 minutes)

# ANCOVA:

- Dependent variable: Change in cortisol concentration (versus baseline)
  at a given time point (for each time point)
- Independent variable: Death vs. survival
- Covariates: Junior vs. senior; Acute vs. non-acute

# Regression:

- Linear regression to determine the effects of covariates (Junior vs. senior; Acute vs. non-acute) on change in cortisol concentration over time
  - Separated into "death" and "survival" groups
  - Change in cortisol concentration will be established using the baseline reading of each participant on each day of the study (time point 1).
- Unpaired t-tests will be used to compare change in cortisol levels between the "death" group and the "survival" group at each time point.

# Measure 2: State-Trait Anxiety Inventory (STAI)

- Analysis will be carried out in the same way as the cortisol measures with the STAI score taking the place of the change in cortisol concentration

## Measure 3: Cognitive appraisal

- Mean cognitive appraisal ratios for each group ("death" and "survival") at each time point will be calculated and subjected to a one-sample t-test to determine whether they are significantly different from 1.
- Unpaired t-tests will be used to compare the mean ratios of the "death" and "survival" groups at each time point.

## **Secondary Outcome 3**: Valence of emotions

Five-point Likert scale

## Repeated measures ANCOVA:

- Dependent variable: Score for each emotion
- Independent variable: Death vs. survival
- Covariates: Junior vs. senior; Acute vs. non-acute
- Time points: Initial and retention

# For all Outcomes:

Relationships between all outcomes (determined by ANCOVA or by Pearson's correlation) will be presented in a matrix table.